CLINICAL TRIAL: NCT01725802
Title: A Phase I/IIa, Single Dose, Single-centre, Randomized, Crossover, Double-blind, Placebo-controlled Study Evaluating Safety, Tolerability and Levodopa Plasma Concentration Following Administration of Subcutaneous Continuously-delivered Levodopa/Carbidopa Solution (ND0612) in PD Patients
Brief Title: A Safety, Tolerability, and Plasma Concentration Study of Levodopa/Carbidopa Subcutaneous Solution (ND0612) in Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND0612/002
Record Dates: First submitted 2012-11-04; First posted 2012-11-14 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence A (Experimental): Period 1. ND0612; Period 2. Placebo
  Interventions: Drug: Levodopa/carbidopa solution for SC administration; Drug: Placebo
- Treatment sequence B (Experimental): Period 1. Placebo; Period 2. ND0612
  Interventions: Drug: Levodopa/carbidopa solution for SC administration; Drug: Placebo

INTERVENTIONS:
Drug: Levodopa/carbidopa solution for SC administration
  Other Names: ND0612
Drug: Placebo
  Other Names: Saline

SUMMARY:
In this Phase I/IIa study, the effect of continuous subcutaneous administration of LD/CD solution (ND0612) on the safety and PK profile of LD will be examined.

DETAILED DESCRIPTION:
Design: single center, double-blind, randomized, placebo-controlled, crossover study.

Study Drug: Subcutaneous (SC), ND0612 (LD/CD solution) or placebo (saline) to be administered via a continuously via the CRONO Five SC pump. A 1-week washout period will apply between the treatments.

Population: Eight (8) PD subjects.

ELIGIBILITY:
Main Inclusion Criteria:

* Men and women with idiopathic Parkinson's disease
* Subjects must experience motor fluctuations associated with LD/CD dosing
* Modified Hoehn and Yahr stage < 5
* Subjects must be taking optimized and stable levodopa/dopa decarboxylase inhibitor therapy
* Women must be postmenopausal, surgically sterilized, or using adequate birth control. Women of childbearing potential must have a negative pregnancy test (serum beta-HCG) at screening.
* Subjects must be age 30 or older.
* Subjects must be willing and able to give informed consent.

Main Exclusion Criteria:

* Subjects with a clinically significant or unstable medical or surgical condition
* Subjects with clinically significant psychiatric illness.
* Pre-menopausal women, not using birth control method.
* Subjects who have taken experimental medications within 60 days prior to baseline.
* Subject who have undergone a neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, transplantation and deep brain stimulation).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-12-16 (Actual); Primary Completion 2013-02-26 (Actual); Study Completion 2013-02-26 (Actual)

PRIMARY OUTCOMES:
Incidence and frequency of adverse events | up to 8 weeks
  1. Incidence and frequency of adverse events
  2. Adverse events reporting related to the ND0612 application, local safety score
Withdrawal rate | 2 days
  Withdrawal rates and discontinuations due to adverse events

SECONDARY OUTCOMES:
LD Half life (t½ ), time of LD plasma concentrations maintained above 1000 ng/ml, trough levels, Cmax, Tmax and AUC | Up to 2 days
  LD PK profile after oral LD dosing administered with or without ND0612:

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel